CLINICAL TRIAL: NCT01304056
Title: How to Study Ventilatory Physiology With the Help of Surface Electromyography (EMG) Recordings
Status: Withdrawn | Type: Observational
Why Stopped: Administrative reasons
Sponsor: Tampere University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: R08175
Record Dates: First submitted 2011-02-24; First posted 2011-02-25 (Estimated); Last update posted 2013-10-09 (Estimated); Status verified 2013-10

CONDITIONS: Ventilatory Physiology
Keywords: Ventilatory physiology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Critically ill patients: Patients that are treated in intensive care unit and given ventilatory therapy.
  Interventions: Device: Ventilatory therapy
- Interventional volunteer group: Healthy volunteers

INTERVENTIONS:
Device: Ventilatory therapy
  Groups: Critically ill patients

SUMMARY:
Respiratory muscles seem to be activating differently in critically ill patients than in healthy persons. Needle electrodes would provide artefact-free signal information about muscle activation. However, needle recordings are an invasive technique which limits its feasibility in clinical setting. Intention of this study is to investigate if surface electromyography could be used to measure recruitment patterns of ventilatory muscles.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age

Exclusion Criteria:

* brain death of injury
* high spinal cord injury
* severe ARDS (static compliance below 40, PFI below 150)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult population > 18 years of age
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-08; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jyrki Tenhunen, MD, PhD, Study Director — Critical Care Medicine Research Group, Tampere University Hospital